CLINICAL TRIAL: NCT05094245
Title: Stellate Gnaglion Block Versus Conventional Therapey in Refractory Bell's Palsy; A Rondomized Single Blind Clinical Trial
Brief Title: Stellate Gnaglion Block in Refractory Bell's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB009999
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Facial Palsy; Neuropathy
Keywords: neuropathy
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate ganglion block (Active Comparator): Patients underwent a stellate-ganglion block at the anterolateral aspect of the C6 vertebra. After local analgesia (lidocaine 2%), a 22-gauge Quincke needle was placed in the anterolateral aspect of the C6 vertebral body. When the needle contacted the bone, it was drawn back 1 mm. 5 mL of 0·5% ropivacaine was subsequently injected next to the stellate ganglion to produce a sympathetic block.The effect of the stellate-ganglion block on the sympathetic nervous system was confirmed by the presence of Horner's syndrome (ie, facial anhydrosis, enophthalmos, ptosis, swelling of the lower eyelid, miosis, and blood-shot conjunctiva), and an increase in the temperature of the right hand of at least 2°F from baseline.
  Interventions: Procedure: Stellate Ganglion Block Group
- Conventional (No Intervention): Mecobalamin Tablets oral Mecobalamin Tablets tid-8

INTERVENTIONS:
Procedure: Stellate Ganglion Block Group — Patients underwent a stellate-ganglion block at the anterolateral aspect of the C6 vertebra. After local analgesia (lidocaine 2%), a 22-gauge Quincke needle was placed in the anterolateral aspect of the C6 vertebral body. When the needle contacted the bone, it was drawn back 1 mm. 5 mL of 0·5% ropivacaine was subsequently injected next to the stellate ganglion to produce a sympathetic block.The effect of the stellate-ganglion block on the sympathetic nervous system was confirmed by the presence of Horner's syndrome (ie, facial anhydrosis, enophthalmos, ptosis, swelling of the lower eyelid, miosis, and blood-shot conjunctiva), and an increase in the temperature of the right hand of at least 2°F from baseline.
  Arms: Stellate ganglion block

SUMMARY:
Idiopathic facial nerve palsy (Bell's palsy) is caused by damage to the facial nerve at any site of the peripheral branches after the facial nucleus.Stellate ganglion block is inteneded to increase blood flow and promotes nerve regeneration.

DETAILED DESCRIPTION:
the conventional systemic corticosteroid treatment for acute peripheral facial nerve palsy in patients can induce hyperglycemia, and an alternative local therapy may be necessary and some time may ve ineffective.

Our purpose in this study is to evaluate therapeutic effects of stellate ganglion block (SGB) on idiopathic persistant facial nerve palsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by clinical and neurological assessment as one-sided idiopathic facial palsy
* Age 18 to 60
* ASA Ⅰ~Ⅲ

Exclusion Criteria:

* diabetic
* coagulation dysfunction
* mental or cognitive dysfunclion
* allergy to injected medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
House Brackmann grading scale | Baseline ,change from baseline House-Brackmann at 7th day,one month,two month, three month
  The House-Brackmann scale is a nerve grading system, It is used to characterize the severity of a facial paralysis patient's symptoms.
  Grade I : 100% functioning Grade VI : 0% function

SECONDARY OUTCOMES:
Likert scale | before intervention , and directly after intervention
  Likert scale (Patients' satisfaction) is typically a five; 1 =strongly dis-satisfied and 5= strongly satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No